CLINICAL TRIAL: NCT05339932
Title: GVSU Skills on Wheels: A Pediatric Manual Wheelchair Skills Training Program
Brief Title: Grand Valley State University (GVSU) Skills on Wheels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Principal Investigator, Lisa Kenyon, Professor, Grand Valley State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-226-H
Record Dates: First submitted 2022-03-30; First posted 2022-04-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Spina Bifida; Cerebral Palsy; Genetic Disease; Spinal Cord Injuries; Gross Motor Development Delay; Motor Skills Disorders
MeSH Terms: conditions — Spinal Dysraphism; Cerebral Palsy; Genetic Diseases, Inborn; Spinal Cord Injuries; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Manual wheelchair skills training (Experimental)
  Interventions: Other: Manual Wheelchair Skills Training

INTERVENTIONS:
Other: Manual Wheelchair Skills Training — The intervention involves manual wheelchair skills training.

SUMMARY:
Manual wheelchairs (MWCs) are widely used by children with physical disabilities, yet many of these children are unable to use their wheelchair independently. Instead, they depend on others to push them. This dependency results in limited opportunities to decide what they want to do and where they want to go, leading to learned helplessness, social isolation, decreased participation, and restricted involvement in physical activities. Furthermore, unsafe MWC use increases the risk of injury, as highlighted by the 44,300 children treated each year in emergency departments for MWC-related injuries. While independent MWC mobility can positively influence quality of life, MWC skills training must also be provided to promote safe, independent MWC use. The effectiveness of MWC training programs for adults is well established, yet the current standard-of-care does not include MWC skills training for children and research regarding the efficacy of pediatric MWC skills training programs is limited. Skills on Wheels seeks to address these gaps and provide pilot data for a future large-scale, multi-site research project involving a randomized controlled trial. Aim 1 is to explore the influence of Skills on Wheels on children's MWC skills and confidence in their MWC use. Aim 2 is to investigate the influence of Skills on Wheels on children's psychosocial skills, social participation, and adaptive behavior.

DETAILED DESCRIPTION:
Manual wheelchairs (MWCs) are widely used by children with physical disabilities, yet many of these children are unable to use their wheelchair independently. Instead, they depend on others to push them. This dependency results in limited opportunities to decide what they want to do and where they want to go, leading to learned helplessness, social isolation, decreased participation, and restricted involvement in physical activities. Furthermore, unsafe MWC use increases the risk of injury, as highlighted by the 44,300 children treated each year in emergency departments for MWC-related injuries. While independent MWC mobility can positively influence quality of life, MWC skills training must also be provided to promote safe, independent MWC use. The effectiveness of MWC training programs for adults is well established, yet the current standard-of-care does not include MWC skills training for children and research regarding the efficacy of pediatric MWC skills training programs is limited. Skills on Wheels seeks to address these gaps and provide pilot data for a future large-scale, multi-site research project involving a randomized controlled trial. The final outcomes and significance of this project are as follows: Aim 1 is to explore the influence of Skills on Wheels on children's MWC skills and confidence in their MWC use and Aim 2 is to investigate the influence of Skills on Wheels on children's psychosocial skills, social participation, and adaptive behavior.

ELIGIBILITY:
Inclusion Criteria:

* 5-17 years of age. NOTE: Participants must be under 18 for the duration of the study.
* Have a condition resulting in difficulties walking.
* Use a manual wheelchair greater than or equal to 25% of the time
* Are able to follow simple instructions per parent report
* Has at least one parent/caregiver who is able to converse in English (as assessed by the PI during interactions over the phone and in person) due to safety concerns.
* Resides in Michigan

Exclusion Criteria:

* Any reason that it would not be safe for the child to participate in manual wheelchair training (as assessed by the PI, a licensed physical therapist)
* The child's manual wheelchair is not safe (as assessed by the PI, a licensed physical therapist)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in manual wheelchair skills performance | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  This outcome will be assessed using the Wheelchair Skills Test (WST) and the Wheelchair Skills Test Questionnaire (WST-Q) scales for performance. These complementary measures were designed to be used together and consist of a 0-3 rating scale for each of the 32 manual wheelchair skills included in these measures.
Change in manual wheelchair skill performance | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  This outcome will be assessed using the Canadian Occupational Performance Measure (COPM) to identify, prioritize,and rate caregiver perceptions of children's performance of manual wheelchair skills and will provide the basis for manual wheelchair skills training intervention. A total of 4-5 occupational performance issues in the area of manual wheelchair skills will be identified and scored on a 1-10 scale for both the caregiver's perception of the child's performance and their satisfaction with the child's performance. This completed with children >8-years-old, if they are able.
Change in manual wheelchair skill confidence | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  This outcome will be assessed using the WheelConPed. This measure consists of a 0-4 rating skill for each of the 33 manual wheelchair use scenarios included in the measure.

SECONDARY OUTCOMES:
Change in behavior | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  This outcome will be measured using the Strengths and Difficulties Questionnaire (SDQ) caregiver questionnaire covering children's behaviors and emotions. The SDQ encompasses 5 subscales: Emotional, Conduct, Hyperactivity/inattention, Peer relationships, and Prosocial behavior. The self-report version will also be completed by children ages 11-17, if they are able.
Change in adaptive skills | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  This outcome will be measured using the Adaptive Behavior Assessment System, 3rd Edition (ABAS), a computer-based caregiver questionnaire to assess children's abilities in 11 adaptive skill areas within 3 domains (conceptual, social, and practical).
Changes in perceptions regarding the manual wheelchair skills intervention | Baseline,pre-intervention and immediately after the conclusion of the 6 week intervention
  Caregivers' perceptions of the manual wheelchair skills intervention will be gathered via a recorded qualitative interview. An interview guide has been developed for this purpose. Children will also participate in a recorded qualitative interview, if able. An interview guide has been developed for this purpose.

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared upon request.